CLINICAL TRIAL: NCT04435431
Title: A Randomized, Double-blind, Placebo-controlled Phase IIB Study Evaluating the Efficacy of Mesdopetam on Daily ON-time Without Troublesome Dyskinesia in Patients With Parkinson's Disease
Brief Title: A Clinical Study of Mesdopetam in Patients With Parkinson's Disease Experiencing Levodopa Induced Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Integrative Research Laboratories AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRL790C005
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — mesdopetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mesdopetam dose 1 (Experimental): Mesdopetam capsule (mg), dose 1, 1 capsule b.i.d. for 84 days.
  Interventions: Drug: Mesdopetam
- Mesdopetam dose 2 (Experimental): Mesdopetam capsule (mg), dose 2, 1 capsule b.i.d. for 84 days.
  Interventions: Drug: Mesdopetam
- Mesdopetam dose 3 (Experimental): Mesdopetam capsule (mg), dose 3, 1 capsule b.i.d. for 84 days.
  Interventions: Drug: Mesdopetam
- Placebo (Placebo Comparator): Placebo capsule, 1 capsule b.i.d. for 84 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesdopetam — Oral use
  Other Names: IRL790
  Arms: Mesdopetam dose 1; Mesdopetam dose 2; Mesdopetam dose 3
Drug: Placebo — Oral use
  Arms: Placebo

SUMMARY:
This is a Phase 2b study investigating the efficacy and safety of mesdopetam as adjunct therapy on daily ON-time without troublesome dyskinesia in patients with Parkinson disease. Mesdopetam is taken for 84 days.

DETAILED DESCRIPTION:
At the screening visit consenting patients will be screened for eligibility according to study specific inclusion/exclusion criteria within 8 weeks before start of Investigational Medicinal Product (IMP) administration. A diary concordance training will be performed and following the screening visit the patient will be asked to self-administer three 24-hour home diaries and to bring the completed diaries to the baseline visit for assessment prior randomization.

At the baseline visit, patients will be randomized to receive one of three doses of mesdopetam (dose 1, dose 2 and dose 3) or placebo b.i.d.

During the first week a dose run-in phase will take place, where all patients allocated to mesdopetam will receive a run-in dose of mesdopetam twice daily and patients allocated to placebo will receive placebo twice daily. At Visit 2, patients will receive mesdopetam dose 1, dose 2 or dose 3 or placebo b.i.d., as randomized and continue the same dose for the rest of the treatment period until end of treatment (EOT). Dose reductions are restricted and the dose can only be reduced once. Dose reductions are permitted from visit 2 (day 9) until visit 3 (day 28), where after the dose should be kept stable until EOT.

The treatment allocation will be double-blind, i.e. it will not be disclosed to the patients, the site staff or the Sponsor.

During the treatment period, changes in disease state and ON phase dyskinesia will be assessed using the Movement Disorder Society revised Unified Parkinson's Disease Rating Scale (MDS-UPDRS), the modified Unified Dyskinesia Rating Scale (UDysRS), i.e. parts 1, 3 and 4, and Clinician's Global Impression of Severity (CGI-S). Furthermore, patients will self-administer three 24-hour home diaries prior to visit 3 (week 4), visit 4 (week 8) and visit 5 (week 12) to assess daily motor function.

Blood samples for pharmacokinetic (PK) analysis will be collected at visit 4 (week 8) and visit 5 (week 12).

Visit 6 (follow-up) will be performed for all patients, including any patients that discontinue the IMP early, 5-8 days after last administration of IMP.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥30 and ≤79 years of age at the time of screening.
2. Signed a current Ethics Committee approved informed consent form (ICF).
3. PD, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria.
4. Minimal amount of 2 hours of levodopa-induced daily "ON-time with troublesome dyskinesia" during waking hours
5. Functional impact of dyskinesias determined as a score of ≥2 as per Question 4.2 of the MDS-UPDRS.
6. On a stable regimen of antiparkinson medications for at least 30 days prior to first home diary completion which must include a levodopa preparation administered 3-8 times/day (excluding nighttime levodopa) and willing to continue the same doses and regimens during study participation. Rescue medications such as Madopar dispersable and Apomorphine injections are allowed if prescribed PRN prior to study entry.
7. Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to first home diary completion and the patient must be willing to continue the same doses and regimens during study participation (this criterion does not apply to medications that are being taken pre-study only on an as-needed basis).
8. Able to complete 24-hour patient home diaries of which two valid diaries must be presented at visit 1.

Exclusion Criteria:

1. History of neurosurgical intervention related to PD (e.g. deep brain stimulation).
2. Treatment with pump delivered antiparkinsonian therapy (i.e. subcutaneous apomorphine or levodopa/carbidopa intestinal infusion).
3. History of seizures within two years prior to screening.
4. History of stroke or transient ischemic attack (TIA) within two years prior to screening.
5. History of cancer within five years prior to screening, with the following exceptions: adequately treated non-melanomatous skin cancers, localized bladder cancer, non metastatic prostate cancer or in situ cervical cancer.
6. Presence of cognitive impairment, as evidenced by a Mini-Mental State Examination (MMSE) score of less than 24 during screening.
7. A Hoehn and Yahr stage of 5.
8. Ongoing treatment with amantadine at time of screening or within 6 weeks prior first home diary completion.
9. Treatment with Inbrija (levodopa inhalation powder) at time of screening or within 4 weeks prior first home diary completion.
10. Any history of a significant heart condition or cardiac arrhythmias within the past 5 years, any repolarisation deficits or any other clinically significant abnormal ECG as judged by the Investigator.
11. Severe or ongoing unstable medical condition including a history of poorly controlled diabetes; obesity associated with metabolic syndrome; uncontrolled hypertension; cerebrovascular disease, or any form of clinically significant cardiac disease, clinically significant symptomatic orthostatic hypotension (a fall and/or a discomfort); clinically significant hepatic disease, severe renal impairment, i.e. creatinine clearance <30 mL/min (stage IV or V).
12. Any history of a neurological disorder other than PD or a psychiatric disorder, including history of Diagnostic and Statistical Manual of Mental Disorders (DSM) IV diagnosed major depression or psychosis. Patients with illusions or hallucinations with no loss of insight will be eligible. Patients with mild depression who are well controlled on a stable dose of an antidepressant medication for at least 4 weeks before screening will be eligible.
13. Enrolment in any other clinical study involving medication, medical devices or surgical procedures, current or within three months prior to screening visit, or previous participation in the present study. Patients enrolled in non-interventional clinical trials will be eligible.
14. Drug and/or alcohol abuse.
15. History of severe drug allergy or hypersensitivity.
16. If female, is pregnant or lactating, or has a positive pregnancy test result pre-dose.
17. Patients unwilling to use two forms of contraception (one of which being a barrier method (see Section 8.1) during the treatment period and 90 days for men and 30 days for women after last IMP dose.
18. Any planned major surgery within the duration of the study.
19. Any other condition or symptoms preventing the patient from entering the study, according to the Investigator's judgement.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Tedroff, Study Director — Integrative Research Laboratories AB (IRLAB)
Locations (44):
- United States (14):
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Collaborative Neuroscience Research (CNS Research), Long Beach, California
  - Parkinson's Disease and Movement Disorders Center of Silicon Valley, Palo Alto, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Avantis Clinical Research, Miami, Florida
  - Elias Research Associates (Allied Biomedical Research Institute), Miami, Florida
  - Pharmax Research of South Florida, Inc., Miami, Florida
  - Life Medical Research Group Corp, Miami Gardens, Florida
  - NeuroStudies.net, LLC, Decatur, Georgia
  - University of Kentucky, Department of Neurology, Lexington, Kentucky
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Inland Northwest Research, Spokane, Washington
- France (6):
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - CHU Dupuytren 1 - Neurologie, Limoges
  - CHU Carémeau, Nîmes
  - CHU de Poitiers, Poitiers
  - CHU Rennes-Pontchaillou, Rennes
  - CHU Charles Nicolle; Service de Neurologie, Rouen
- Israel (5):
  - Rambam Health Care Campus, Department of Neurology, Haifa
  - Hadassah University Hospital-Ein Kerem, Department of Neurology, Jerusalem
  - Rabin Medical Centre - Beilinson Hospital, Department of Neurology, Petah Tikva
  - The Chaim Sheba Medical Centre, Department of Neurology, Ramat Gan
  - Tel Aviv Sourasky Medical Centre; Movement Disorders Unit, Tel Aviv
- Italy (5):
  - IRCCS - Ospedale "San Martino", Genova
  - Azienda Ospedaliera di Padova, Padua
  - IRCCS San Raffaele Pisana, Roma
  - Fondazione Policlinico Gemelli IRCCS, Roma
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Clinica Neurologica, Salerno
- Poland (10):
  - Centrum Medyczne Neuromed, Bydgoszcz
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Centrum Medyczne PLEJADY, Krakow
  - Specjalistyczne Gabinety Sp z o.o., Krakow
  - Krakowska Akademia Neurologii, Krakow
  - Instytut Zdrowia, Oświęcim
  - Neuro-Care, Siemianowice Śląskie
  - Centrum Medyczne NeuroProtect, Warsaw
  - Next Stage sp.z o.o., Warsaw
  - ClinHouse Centrum Medyczne, Zabrze
- Serbia (4):
  - Clinical Hospital Center Zvezdara, Clinical department of Neurology, Belgrade
  - University Clinical Center of Serbia, Clinic for Neurology, Belgrade
  - University Clinical Center Kragujevac, Clinic for Neurology (Site 601), Kragujevac
  - University Clinical Center Kragujevac, Clinic for Neurology (Site 602), Kragujevac

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becanovic K, Vittoria de Donno M, Sousa VC, Tedroff J, Svenningsson P. Effects of a Novel Psychomotor Stabilizer, IRL790, on Biochemical Measures of Synaptic Markers and Neurotransmission. J Pharmacol Exp Ther. 2020 Jul;374(1):126-133. doi: 10.1124/jpet.119.264754. Epub 2020 May 1. PMID 32358047
- [Background] Waters S, Sonesson C, Svensson P, Tedroff J, Carta M, Ljung E, Gunnergren J, Edling M, Svanberg B, Fagerberg A, Kullingsjo J, Hjorth S, Waters N. Preclinical Pharmacology of [2-(3-Fluoro-5-Methanesulfonyl-phenoxy)Ethyl](Propyl)amine (IRL790), a Novel Dopamine Transmission Modulator for the Treatment of Motor and Psychiatric Complications in Parkinson Disease. J Pharmacol Exp Ther. 2020 Jul;374(1):113-125. doi: 10.1124/jpet.119.264226. Epub 2020 May 1. PMID 32358046
- [Background] Svenningsson P, Johansson A, Nyholm D, Tsitsi P, Hansson F, Sonesson C, Tedroff J. Safety and tolerability of IRL790 in Parkinson's disease with levodopa-induced dyskinesia-a phase 1b trial. NPJ Parkinsons Dis. 2018 Dec 6;4:35. doi: 10.1038/s41531-018-0071-3. eCollection 2018. PMID 30534585

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesdopetam 2.5 mg: Mesdopetam capsule (2.5 mg), 1 capsule b.i.d. for 84 days.
  Mesdopetam: Oral use
- Mesdopetam 5 mg: Mesdopetam capsule (5 mg), 1 capsule b.i.d. for 84 days.
  Mesdopetam: Oral use
- Mesdopetam 7.5 mg: Mesdopetam capsule (7.5 mg), 1 capsule b.i.d. for 84 days.
  Mesdopetam: Oral use
Period: Overall Study
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo
Started | 40 | 38 | 38 | 39
Completed | 32 | 31 | 29 | 33
Not Completed | 8 | 7 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo | Total
Number analyzed (Participants) | 40 | 38 | 38 | 39 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 17 | 16 | 65
  >=65 years | 23 | 23 | 21 | 23 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (9.3) | 64.9 (9.6) | 65.0 (10.2) | 64.5 (8.5) | 64.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 17 | 25 | 73
  Male | 26 | 21 | 21 | 14 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 5 | 6 | 15
  Not Hispanic or Latino | 38 | 36 | 33 | 33 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 3
  White | 40 | 35 | 36 | 39 | 150
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 11 | 8 | 36
  Poland | 18 | 15 | 12 | 17 | 62
  Italy | 4 | 6 | 3 | 2 | 15
  Israel | 1 | 2 | 3 | 1 | 7
  France | 5 | 4 | 5 | 6 | 20
  Serbia | 3 | 3 | 4 | 5 | 15
Height at Screening [Mean (Standard Deviation); unit: cm] | 167.8 (7.6) | 167.0 (8.8) | 167.8 (8.5) | 165.7 (9.3) | 167.1 (8.5)
Weight at Screening [Mean (Standard Deviation); unit: kg] | 76.9 (15.0) | 73.1 (14.8) | 73.1 (13.7) | 70.3 (17.3) | 73.4 (15.3)
BMI at Screening [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.3) | 26.1 (4.6) | 26.0 (5.0) | 25.6 (6.1) | 26.2 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Hours of ON-time Without Troublesome Dyskinesia With Mesdopetam Compared to Placebo as Assessed With 24-hour Patient Home Diaries From Baseline to End of Treatment.
Description: This is a self-administered diary where patients assess their motor state every half hour during 24 hours. ON time without troublesome dyskinesia measures time when the medication is working without causing troublesome dyskinesia.
Time Frame: Baseline to end of treatment (week 12)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: hours per day
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo
Number analyzed (Participants) | 35 | 35 | 33 | 37
hours per day | 1.211 (0.4895) | 1.737 (0.5028) | 2.233 (0.5278) | 1.985 (0.4776)

2. Secondary Outcome: Change From Baseline in Mean Score of ON-phase Dyskinesia Assessed With the Sum Score of the Modified Unified Dyskinesia Rating Scale (UDysRS), Parts 1, 3 and 4, With Mesdopetam Compared to Placebo.
Description: The scoring range is 0-88, where higher score means more dyskinesia.
Time Frame: Baseline to end of treatment (week 12)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Units on the scale
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo
Number analyzed (Participants) | 35 | 35 | 33 | 37
Units on the scale | -11.5 (1.90) | -9.3 (1.92) | -12.0 (2.00) | -5.8 (1.87)

3. Secondary Outcome: Change From Baseline in Mean Score of Disability Associated With ON-phase Dyskinesia Assessed With the Sum Score of Parts 1b and 4 of the Unified Dyskinesia Rating Scale (UDysRS), With Mesdopetam Compared to Placebo.
Description: The scoring range is 0-60, where higher score means more disability associated with dyskinesia.
Time Frame: Baseline to end of treatment (week 12)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Units on the scale
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo
Number analyzed (Participants) | 35 | 35 | 33 | 37
Units on the scale | -6.3 (1.27) | -5.8 (1.28) | -7.2 (1.33) | -3.7 (1.24)

4. Secondary Outcome: Change From Baseline in Mean Score of Motor Symptoms of PD Assessed With MDS-UPDRS Total Score of Part 2 (M-EDL) (With Mesdopetam Compared to Placebo)
Description: This scale is a patient reported outcome measure assessing motor aspects of experiences of daily living. Minimum score is 0 and maximum score is 52. A higher score means more Parkinson's disease motor symptoms.
Time Frame: Baseline to end of treatment (week 12)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Total Score
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo
Number analyzed (Participants) | 35 | 35 | 33 | 37
Total Score | -0.9 (0.78) | -0.7 (0.79) | 0.0 (0.82) | 0.0 (0.77)

5. Secondary Outcome: Change From Baseline in Average Daily Hours of OFF-time (With Mesdopetam Compared to Placebo).
Description: This is a self-administered diary where patients assess their motor state every half hour during 24 hours. OFF time means time means daily time spent when the medication is not working.
Time Frame: Baseline to end of treatment (week 12)
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: hours per day
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo
Number analyzed (Participants) | 35 | 35 | 33 | 37
hours per day | -0.029 (0.3431) | -0.324 (0.3522) | -0.768 (0.3689) | -0.069 (0.3352)

ADVERSE EVENTS:
Time Frame: Collection of AEs started after the patient signed the ICF (Screening visit) and continued until the last follow-up assessment (End of Study visit/Early Withdrawal visit) in total up to 21 weeks.
Arm/Group | Mesdopetam 2.5 mg | Mesdopetam 5 mg | Mesdopetam 7.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/38 | 1/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/38 | 2/38 | 3/39
Other Adverse Events (participants affected / at risk) | 9/40 | 7/38 | 6/38 | 9/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesdopetam 2.5 mg (N=40) | Mesdopetam 5 mg (N=38) | Mesdopetam 7.5 mg (N=38) | Placebo (N=39)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhytmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesdopetam 2.5 mg (N=40) | Mesdopetam 5 mg (N=38) | Mesdopetam 7.5 mg (N=38) | Placebo (N=39)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5) | 2 (5) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (2) | 2 (2) | 1 (2) | 4 (4)
Dyskinesia (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 2 (5) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Protection of potential intellectual property of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04435431/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04435431/SAP_001.pdf